CLINICAL TRIAL: NCT01210040
Title: Malaria Risk Prior to and During Early Pregnancy in Nulliparous Women Receiving Long-term Weekly Iron and Folic Acid Supplementation (WIFS): a Non-inferiority Randomized Controlled Trial
Brief Title: Long-term Iron Supplements and Malaria Risk in Early Pregnancy: a Randomized Controlled Trial
Acronym: PALUFER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Institute of Tropical Medicine, Belgium (Other); University of Manchester (Other); Institut de Recherche en Sciences de la Sante-Direction Regionale de l'Ouest (Other Government); Centre Muraz (Other); National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 10.55; 1U01HD061234-01A1 (NIH)
Record Dates: First submitted 2010-09-27; First posted 2010-09-28 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Malaria
Keywords: Pregnancy; Iron deficiency; Iron supplementation; Burkina Faso
MeSH Terms: conditions — Malaria; Iron Deficiencies | interventions — Folic Acid; Iron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Folic Acid (Active Comparator): 2.8mg of Folic Acid given weekly
  Interventions: Dietary Supplement: Folic Acid
- Folic Acid and Iron (Experimental): 2.8mg Folic Acid and 60mg Iron given weekly
  Interventions: Dietary Supplement: Folic Acid and Iron

INTERVENTIONS:
Dietary Supplement: Folic Acid — 2.8mg
  Arms: Folic Acid
Dietary Supplement: Folic Acid and Iron — 60mg Iron and 2.8mg Folic Acid
  Arms: Folic Acid and Iron

SUMMARY:
A randomized double-blind controlled trial will be carried out in which young, nulliparous (having never given birth) women will be randomly assigned to receive weekly supplementation with either iron and folic acid or folic acid alone. Women will be followed-up weekly up to 18 months. Women who become pregnant will be followed-up until delivery. Malaria risk in both groups will be compared by assessing the prevalence of peripheral parasitaemia at the first antenatal clinic visit for pregnant women and at the end of the first malaria transmission season for non-pregnant women. The incidence of clinical malaria will be assessed by active and passive case detection throughout the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Female
* At least 15 and less than 25 years old at enrolment
* Never given birth
* Resident within the Demographic Surveillance System (DSS) area
* Willing to adhere to the study requirements (including weekly observed drug intake)
* Provision of written informed consent (if non emancipated minor by guardian/parent with minor's assent

Exclusion Criteria:

* No menses for >3 months and/or palpable uterus or positive pregnancy test if history unclear
* Concurrent enrolment in another study
* Intention to move out of the study area for more than 2 months within the next 18 months
* Any significant illness at the time of screening that requires hospitalization, including clinical signs of severe anaemia (conjunctival or mucosal pallor, tachycardia, respiratory distress)
* History or presence of major clinical disease likely to influence pregnancy outcome (sickle cell disease, diabetes mellitus, severe renal or heart disease, open tuberculosis, epilepsy)

Ages: 15 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1959 (Actual)
Dates: Start 2011-04; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of peripheral parasitaemia at first antenatal clinic visit (13-16 weeks gestation) | Nov 2013
  Completed

SECONDARY OUTCOMES:
a) In the pregnant cohort: Prevalence of iron deficiency at first antenatal visit | Sept 2013
  Completed
a) In the pregnant cohort: Prevalence of anaemia at first antenatal clinic visit | Sept 2013
  Completed
a) In the pregnant cohort: Incidence of clinical malaria during the first and subsequent trimesters | Jan 2014
  Completed
a) In the pregnant cohort: Incidence of adverse pregnancy outcomes | Jan 2014
  Completed
a) In the pregnant cohort: Mean birth weight and prevalence of low birth weight (<2500g) | Jan 2014
  Completed
a) In the pregnant cohort: Mean gestational age at delivery | Jan 2014
  Completed
a) In the pregnant cohort: Prevalence of placental malaria | Jan 2014
  Completed
a) In the non-pregnant cohort: Prevalence of peripheral parasitaemia during the first rainy season after at least six months of supplementation | Nov 2012
  Completed
a) In the non-pregnant cohort: Incidence of clinical malaria | Nov 2013
  Completed
a) In the non-pregnant cohort: Incidence of gastrointestinal adverse events | Nov 2013
  Completed
a) In the non-pregnant cohort: Prevalence of iron deficiency after at least 18 months supplementation | Nov 2013
  Completed
a) In the non-pregnant cohort: Prevalence of anaemia after at least 18 months supplementation | Nov 2013
  Completed
a) In the non-pregnant cohort: Adherence to supplementation | Nov 2013
  Completed
a) In the non-pregnant cohort: Acceptability of weekly supplementation | June 2013
  Completed
In the non-pregnant cohort: Prevalence of bacterial vaginosis at end assessment | Nov 2013
  Completed
a) In the non-pregnant cohort: Prevalence of bacterial vaginosis at end assessment | Nov 2013
  Completed
a) In the non-pregnant cohort: Prevalence of bacterial vaginosis at first antenatal visit | Nov 2013
  Completed
a) In the non-pregnant cohort: Prevalence of iron deficiency at key study visits | Nov 2013
  Completed
a) In the non-pregnant cohort: Prevalence of peripheral parasitaemia at end assessment | Nov 2013
  Completed

CONTACTS AND LOCATIONS:
Overall Officials: Bernard J BRABIN, Professor, Study Director — Liverpool School of Tropical Medicine; Sabine GIES, MD, MTropMed, PhD, Principal Investigator — Clinical Research Unit Nanoro (CRUN)
Locations (1):
- Institute de Recherche en Sciences de la Sante, Direction Regionale de l'Ouest (IRSS-DRO) - / Centre Muraz, Bobo-Dioulasso, Burkina Faso

REFERENCES:
- [Derived] Brabin B, Tinto H, Roberts SA. Testing an infection model to explain excess risk of preterm birth with long-term iron supplementation in a malaria endemic area. Malar J. 2019 Nov 26;18(1):374. doi: 10.1186/s12936-019-3013-6. PMID 31771607
- [Derived] Brabin B, Gies S, Roberts SA, Diallo S, Lompo OM, Kazienga A, Brabin L, Ouedraogo S, Tinto H. Excess risk of preterm birth with periconceptional iron supplementation in a malaria endemic area: analysis of secondary data on birth outcomes in a double blind randomized controlled safety trial in Burkina Faso. Malar J. 2019 May 6;18(1):161. doi: 10.1186/s12936-019-2797-8. PMID 31060615
- [Derived] Diallo S, Roberts SA, Gies S, Rouamba T, Swinkels DW, Geurts-Moespot AJ, Ouedraogo S, Ouedraogo GA, Tinto H, Brabin BJ. Malaria early in the first pregnancy: Potential impact of iron status. Clin Nutr. 2020 Jan;39(1):204-214. doi: 10.1016/j.clnu.2019.01.016. Epub 2019 Jan 26. PMID 30737046
- [Derived] Gies S, Diallo S, Roberts SA, Kazienga A, Powney M, Brabin L, Ouedraogo S, Swinkels DW, Geurts-Moespot AJ, Claeys Y, D'Alessandro U, Tinto H, Faragher B, Brabin B. Effects of Weekly Iron and Folic Acid Supplements on Malaria Risk in Nulliparous Women in Burkina Faso: A Periconceptional, Double-Blind, Randomized Controlled Noninferiority Trial. J Infect Dis. 2018 Aug 24;218(7):1099-1109. doi: 10.1093/infdis/jiy257. PMID 29733403
- [Derived] Compaore A, Gies S, Brabin B, Tinto H, Brabin L. Community approval required for periconceptional adolescent adherence to weekly iron and/or folic acid supplementation: a qualitative study in rural Burkina Faso. Reprod Health. 2018 Mar 14;15(1):48. doi: 10.1186/s12978-018-0490-y. PMID 29540225
- [Derived] Brabin L, Roberts SA, Gies S, Nelson A, Diallo S, Stewart CJ, Kazienga A, Birtles J, Ouedraogo S, Claeys Y, Tinto H, d'Alessandro U, Faragher EB, Brabin B. Effects of long-term weekly iron and folic acid supplementation on lower genital tract infection - a double blind, randomised controlled trial in Burkina Faso. BMC Med. 2017 Nov 23;15(1):206. doi: 10.1186/s12916-017-0967-5. PMID 29166928